CLINICAL TRIAL: NCT04260425
Title: A Randomized Controlled Pilot Study Evaluating the Effect of Oat Polyphenols on Post-prandial Glucose Response in Healthy Adults.
Brief Title: A Pilot Study Evaluating Oat Polyphenols on Post-prandial Glucose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Dylan MacKay. PhD, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HS23437 (B2019:114)
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Blood Glucose
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High then low avenanthramides content oats (Experimental): This arm will receive the high avenanthramides content oatmeal at the first session and the low avenanthramides content oatmeal at the second session. Sessions will be at least 5 days apart.
  Interventions: Other: Serving of oatmeal made from low avenanthramides oats and water; Other: Serving of oatmeal made from high avenanthramides oats and water
- Low then high avenanthramides content oats (Experimental): This arm will receive the low avenanthramides content oatmeal at the first session and the high avenanthramides content oatmeal at the second session. Sessions will be at least 5 days apart.
  Interventions: Other: Serving of oatmeal made from low avenanthramides oats and water; Other: Serving of oatmeal made from high avenanthramides oats and water

INTERVENTIONS:
Other: Serving of oatmeal made from low avenanthramides oats and water — One serving size (40 grams dry weight) of low avenanthramides oats flakes will be used to make oatmeal. One cup of water and a dash of salt (0.72 g) will be added into the treatment and microwaved on high for 3 minutes. It will be stirred before serving. Ingredients and cooking time will be consistently maintained throughout.
Other: Serving of oatmeal made from high avenanthramides oats and water — One serving size (40 grams dry weight) of high avenanthramides oats flakes will be used to make oatmeal. One cup of water and a dash of salt (0.72 g) will be added into the treatment and microwaved on high for 3 minutes. It will be stirred before serving. Ingredients and cooking time will be consistently maintained throughout.

SUMMARY:
The trial will use a two period acute double-blind cross-over design to compare the effects of a serving of oatmeal containing high or low amounts of avenanthramides (AV) on post-prandial blood glucose response in healthy adults.

DETAILED DESCRIPTION:
The clinical trial will follow a two period acute double-blind cross-over design. It will take place at Richardson Centre for Functional Food and Nutraceuticals (RCFFN) at University of Manitoba, Winnipeg, Canada.

The trial will recruit healthy adult participants. Participants will consent to participate in two acute feeding sessions. Participants will be randomized to either control (low avenanthramides) then treatment (high avenanthramides) or treatment then control. Participants will arrive at the study center fasted between 8 and 10:30 am on the session days. They will be provided either the study treatment or control product based on randomization sequence for their first study visit. Baseline blood glucose (0 min) will be measured in duplicate via finger stick blood sample right before their first bite of the treatment product, and at 15, 30, 45, 60, 90 and 120 mins after baseline. The timer will be started when they take their first bite. During the second visit participant will consume the other treatment based on the randomization (the oatmeal that they didn't receive in their first visit and follow exactly the same procedure as the first visit). There will be a minimum of 5 days between sessions. Female participants will be scheduled during the luteal phase of their menstruation cycle. There will be a maximum of 8 weeks between the two sessions, therefore, participants will finish the both sessions within an 8 week period.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or female between 18-50 years old
* BMI range in between 18.9-29.9 kg/m^2
* Fasting glucose <5.6 mmol/L
* Usually eat breakfast
* In the Investigator's opinion is able and willing to comply with all trial requirements

Exclusion Criteria:

* Fasting glucose ≥ 5.6 mmol/L or <3.5 mmol/L
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Participants who indicate that they could not finish consuming the study treatments within 10 minutes
* Use of medication or supplements that may influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of screening visit
* History of disordered eating, AIDS, hepatitis, a history of clinically important endocrine (including Type I and Type II diabetes mellitus), cardiovascular (including but not limit to atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders
* Intolerance or allergic reaction to oats
* Existing restrictive dietary habits (such a vegan, low carbohydrate or keto)
* Uncontrolled hypertension
* History of cancer within the last two years (except for non-melanoma skin cancer)
* Recent history of (within 12 month of screening) or current strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week, (1 drink = 12oz of beer, 5oz of wine or 1.5oz distilled spirits)
* Body weight change over 3.5kg within the past 3 months
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks
* Had significant physical trauma or major surgery in the past 3 month or had trauma or major surgery in the past 3 month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
post-prandial glucose response | Area under the curve from 0,15, 30, 45, 60, 90 and 120 minutes
  2 hour area under the curve of post-prandial glucose response to the interventions in mmol/L*min^2

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Mackay, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Center for Food Technology and Research, Winnipeg, Manitoba, Canada